CLINICAL TRIAL: NCT00492245
Title: Phototherapeutic Keratectomy With Mitomycin C in Adenoviral Infiltrates
Brief Title: Phototherapeutic Keratectomy (PTK) With Mitomycin in Adenoviral Opacities
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Federal University of São Paulo (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CEP0075/06
Record Dates: First submitted 2007-06-26; First posted 2007-06-27 (Estimated); Last update posted 2008-08-04 (Estimated); Status verified 2008-07

CONDITIONS: Keratitis; Corneal Opacity
Keywords: PTK; corneal opacity; mitomycin
MeSH Terms: conditions — Keratitis; Corneal Opacity | interventions — Mitomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: PTK with mitomycin in Adenoviral Opacities

SUMMARY:
The present study was designed to evaluate the treatment of adenoviral corneal opacities with PTK and mitomycin C.

DETAILED DESCRIPTION:
Epidemic keratoconjunctivitis is a very common disease, some patients developed a complication after the infection wich is corneal infiltration. Topical treatment sometimes helps to avoid loss of visual acuity. Therefore recurrence of the opacities after topical drops is observed. When corneal fibrosis occur is difficult to achieve visual rehabilitation with topical approach. This study evaluate pre and postoperative data of patients with subepithelial fibrosis caused by adenoviral infiltrates submitted to phototherapeutic keratectomy (PTK) using mitomycin C.

ELIGIBILITY:
Inclusion Criteria:

* visual acuity worse than 20/40, caused by central subepithelial fibrosis

Exclusion Criteria:

* pregnancy, age less than 18 years-old or more than 80 years-old.
* diabetes, autoimmune diseases, corneal thickness less tha 400 micron.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2006-04; Primary Completion 2008-05; Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
Refractive data, visual acuity, slit lamp findings, subjective evaluation, topography patterns, pachymetry measurements. | one year

SECONDARY OUTCOMES:
wavefront analysis, anterior segment tomography data, corneal biomechanics data. | one year

CONTACTS AND LOCATIONS:
Overall Officials: Ester S Yamazaki, MD, Principal Investigator — Federal University of Sao Paulo - Brazil; Mauro S Campos, MD, Study Chair — Federal University of Sao Paulo - Brazil
Locations (1):
- Federal University of Sao Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Fagerholm P. Phototherapeutic keratectomy: 12 years of experience. Acta Ophthalmol Scand. 2003 Feb;81(1):19-32. doi: 10.1034/j.1600-0420.2003.00015.x. PMID 12631015
- [Background] Porges Y, Ben-Haim O, Hirsh A, Levinger S. Phototherapeutic keratectomy with mitomycin C for corneal haze following photorefractive keratectomy for myopia. J Refract Surg. 2003 Jan-Feb;19(1):40-3. doi: 10.3928/1081-597X-20030101-08. PMID 12553604
- [Background] Khurana RN, Li Y, Tang M, Lai MM, Huang D. High-speed optical coherence tomography of corneal opacities. Ophthalmology. 2007 Jul;114(7):1278-85. doi: 10.1016/j.ophtha.2006.10.033. Epub 2007 Feb 20. PMID 17307254
- [Derived] Yamazaki ES, Ferraz CA, Hazarbassanov RM, Allemann N, Campos M. Phototherapeutic keratectomy for the treatment of corneal opacities after epidemic keratoconjunctivitis. Am J Ophthalmol. 2011 Jan;151(1):35-43.e1. doi: 10.1016/j.ajo.2010.07.028. Epub 2010 Nov 24. PMID 21109229